CLINICAL TRIAL: NCT04081922
Title: Postoperative Analgesia With Erector Spinae Plane Block After Pectus Excavatum Repair in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1907-087-1049
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional analgesia using erector spinae plane block (Experimental): After pectus excavatum is done, intravenous patient controlled analgesia device with fentanyl is connected. Then, regional analgesia is performed for additional analgesia; ultrasound guided erector spinae plane block is performed using 0.25% ropivacaine (total 1 ml/kg) bilaterally. Plasma concentration of ropivacaine at baseline, and 5, 10, 20, 30, 60, 120 minutes after ropivacaine injection will be measured.
  Interventions: Procedure: Erector spinae plane block
- Control (No Intervention): After pectus excavatum is done, intravenous patient controlled analgesia device with fentanyl is connected. No regional block is performed.

INTERVENTIONS:
Procedure: Erector spinae plane block — Using ultrasound, place the needle in the erector spinae fascia plane at T7-8 level. Then, 0.25% ropivacaine 0.5 ml is injected to confirm the needle location. After checking the location, 0.25% ropivacaine 0.5 ml/kg is administered. This procedure is repeated at contralateral side.
  Arms: Regional analgesia using erector spinae plane block

SUMMARY:
The purpose of this study is to evaluate the efficacy of erector spinae plane (ESP) block in children after pectus excavatum repair (nuss procedure).

ELIGIBILITY:
Inclusion Criteria:

* 30 children aged between 3 and 7 years who undergo Nuss bar insertion due to Pectus excavatum

Exclusion Criteria:

* Allergy to opioid
* Allergy to local anesthetics
* Disease in heart, lung, kidney, and liver
* Coagulation disorder
* Disease in central and peripheral nervous system

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | 1 hour after surgery
  The Face, Legs, Activity, Cry, Consolability (FLACC) scale is used. FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
Fentanyl dosage (mcg/kg) | until hospital discharge (postoperative day 3)
  Total dosage of fentanyl used postoperatively via patient controlled analgesia (mcg/kg)
Dose of rescue analgesics (mg/kg) | until hospital discharge (postoperative day 3
  If additional analgesics are required due to uncontrolled pain, intravnous acetaminophen and ketocin can be administered.
Plasma concentration of ropivacaine | 5, 10, 20, 30, 60, 120 minutes after injection
  Plasma concentration of ropivacaine after injection

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided